CLINICAL TRIAL: NCT00155597
Title: The Outcome and Cost Analysis of Home-care Physical Therapy for Postoperative Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jau-Yih Tsauo, School and Graduate Institude of Physical Therapy, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24368
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-12

CONDITIONS: Hip Fractures
Keywords: physical therapy; post surgery
MeSH Terms: conditions — Hip Fractures

INTERVENTIONS:
Behavioral: home physical therapy

SUMMARY:
The aims of this study are:

1. To develop a disease-specific questionnaire for hip fractures.
2. To find the influences of physical therapy (PT) on patients' function and health-related quality of life (HRQL).
3. To estimate the quality adjusted life years (QALY) of cases of hip fracture with or without the PT program by a quality-adjusted survival (QAS) method.
4. To perform cost effectiveness analysis (CEA) to evaluate the effectiveness of PT and as a base to compare it with other health intervention programs.

At the beginning of the study, the investigators will develop the disease-specific questionnaire for hip fractures. Cases of patients with hip fractures hospitalized in orthopedic wards of the National Taiwan University Hospital (NTUH) and Chung-Hsing Hospital of Taipei from August 1, 1989 to July 31, 1999 are the study population during the first year of this study. According to their receiving PT or not during hospitalization, the patients are assigned to a PT or non-PT group. The identification (ID) numbers will be matched with the death certificate file of the Department of Health to verify the survival status. Furthermore, 30 cases per group per year will be randomly sampled to interview their HRQL and evaluate their function with the disease-specific questionnaire for hip fractures. Combining the survival function and HRQL, the QALY could be estimated. Cases of hip fracture admitted to the orthopedic ward of NTUH and receiving a PT program from January 1, 2000 will be the second-year study population in this study. They will be randomly assigned to a group of follow-up PT (group I) or non-follow-up PT (group II). The patients assigned to group I will have a 4-time PT evaluation and treatment at home after discharge from the hospital (1 week, 1 month, 3 months and 6 months after discharge). All patients will be evaluated at discharge, 1 month, 6 months, and 1 year after discharge to follow their survival status, functional status and HRQL. The expected results of this study will be to develop the disease-specific questionnaire for hip fractures, to show the functional outcomes of cases of hip fracture, and to estimate the QALY of them.

DETAILED DESCRIPTION:
Hip fracture from fall is the most important cause of disability of the aged. Most of the victims receive surgery (internal fixation or arthroplasty) as the primary treatment. However, during the hospitalization of post-surgery, not all the patients receive physical therapy (PT). The program of PT during hospitalization and after discharge affects the functional recovery and the health-related quality of life (HRQL) significantly in our knowledge. Therefore, the aims of this study are:

1. To develop the disease-specific questionnaire for hip fracture.
2. To find the influences of PT on patients' function and HRQL.
3. To estimate the QALY of cases of hip fracture with or without PT program by quality-adjusted survival (QAS) method.
4. To perform CEA to evaluate the effectiveness of PT and as a base to compare with other health intervention program.

At the beginning of the study, we will develop the disease-specific questionnaire for hip fracture. And, cases of hip fracture hospitalized in orthopedic wards of National Taiwan University Hospital (NTUH) and Chung-Hsing Hospital of Taipei from August 1, 1989 to July 31, 1999 are the study population of the first year in this study. According to their receiving PT or not during hospitalization, the patients are assigned to PT or non-PT group. Basic data such as ID number, age, sex, comorbidity, pre-injury physical status, operation date, operation type, length of hospitalization, complication, are extracted from their charts. The identification (ID) numbers will be matched with the death certificate file of the Department of Health to make sure the survival status. Furthermore, 30 cases per group per year will be randomly sampled to interview their HRQL and evaluate their function with the disease-specific questionnaire for hip fracture. Combining the survival function and HRQL, the QALY could be estimated. Cases of hip fracture admit to the orthopedic ward of NTUH and receive PT program from Jan. 1, 2000 will be the second-year study population in this study. They will be randomly assigned to group of follow-up PT (group I) or non-follow-up PT (group II). The patients assigned to group I will have 4-time PT evaluation and treatment at home after discharge from hospital (1 week, 1-month, 3-month and 6-month after discharge). All patients will be evaluated at discharge, 1-month, 6-month, and 1-year after discharge to follow their survival status, functional status and HRQL. The patients younger than 65 years old will be further evaluated for their working capacity at the last evaluation. In the third year of this study, medical cost and estimated QALY will be collected to perform the CEA for the effectiveness of PT program during hospitalization and after discharge.

The expected results of this study will be to develop the disease-specific questionnaire for hip fracture, to show the functional outcome of cases with hip fracture, to estimate the QALY of them and to perform a CEA to demonstrate the effectiveness of PT.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture, post surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-08; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life, Harris score, walking velocity, strength

CONTACTS AND LOCATIONS:
Overall Officials: J Y Tsauo, PhD, Study Director — Grad School of PT, College of Medicine, NTU